CLINICAL TRIAL: NCT05315999
Title: Protreat-Trial: Prophylactic Antiemetic Treatment of Opioid-induced Nausea and Vomiting (OINV) in Palliative Care: a Randomized Controlled Phase II Feasibility Trial
Brief Title: Protreat-Trial: Prophylactic Antiemetic Treatment of Opioid-induced Nausea and Vomiting (OINV) in Palliative Care
Acronym: ProTreat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gerhild Becker (Other)
Responsible Party: Sponsor-Investigator, Gerhild Becker, Prof. Dr. med., University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P003161
Record Dates: First submitted 2022-03-02; First posted 2022-04-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-12

CONDITIONS: Nausea; Vomiting; Pain; Advanced Cancer
MeSH Terms: conditions — Nausea; Vomiting; Pain | interventions — Palonosetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palonosetron Hydrochloride (Experimental): Palonosetron (500µg): single dose per os 1-2 hours before the start of opioid-therapy (WHO II & III)
  Interventions: Drug: Palonosetron Hydrochloride
- Placebo (Placebo Comparator): Placebo: single dose per os 1-2 hours before the start of opioid-therapy (WHO II & III)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Palonosetron Hydrochloride — Palonosetron (500µg): single dose per os 1-2 hours before the start of opioid-therapy (WHO II & III)
  Arms: Palonosetron Hydrochloride
Drug: Placebo — Placebo: single dose per os 1-2 hours before the start of opioid-therapy (WHO II & III)
  Arms: Placebo

SUMMARY:
Palliative cancer patients with tumor pain often suffer from nausea and vomiting when starting pain therapy with opioids. The objective of the clinical pilot trial is to evaluate the efficacy and tolerability of palonosetron in the prophylactic treatment of opioid-induced nausea and vomiting.

DETAILED DESCRIPTION:
Pain is one of the most common and debilitating symptoms in patients with advanced cancer and opioids are the main stay of treatment for cancer pain. However, initiation of opioid-therapy is frequently hindered by OINV. OINV is a highly distressing symptom and can affect medication compliance, enteral absorption, and quality of life.This Phase II feasibility study is conducted to assess the feasibility of the prophylactic antiemetic treatment of OINV with palonosetron in comparison to placebo. The objective is to investigate the feasibility of patient recruitment and implementation of the study design as well as to obtain an initial estimate of the antiemetic efficacy and safety of prophylactic treatment of OINV with palonosetron compared to placebo. A total of 30 palliative patients starting an opioid-therapy (WHO II & III) for cancer pain will be randomly assigned to receive either a single dose of placebo or palonosetron. Safety and efficiency assessment are based on patient reports regarding OINV, pain and safety parameters during the following 6 days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years
2. Opioid naïve (no opioids intake within last 72 hours) patients in whom opioid therapy (WHO II & III) is started to treat cancer pain;
3. Palliative (not curable) cancer pain patients;
4. Patients must have a score for nausea on a 0-10 numeric rating scale (NRS) < 3 at screening visit;
5. Written informed consent obtained according to international guidelines and local laws;
6. Ability of patient to understand nature, importance, and individual consequences of clinical trial;
7. Patients must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patient's death is imminent (judged by the "surprise" question of the treating physician or nurse: "Would you be surprised if this patient died within the next 7 days?"); If the answer is "no", trial subject cannot participate;
2. Participation in the trial considered inappropriate based on the patient's physical, social, psychological, or spiritual condition (judgement of treating physician or nurse);
3. Patients receiving antiemetic treatment within the last 72 h before study treatment period
4. Patients if they are known to start a treatment causing acute nausea and/or emesis during study period
5. Patients with contraindications or hypersensitivity to opioids or palonosetron, fructose, soya, lactose or peanut intolerance;
6. Patients unable to take oral medications or patients receiving medication via PEG-tube;
7. Patients undergoing dialyses treatment;
8. Known or persistent abuse of medication, drugs, or alcohol;
9. Current or planned pregnancy, nursing period;
10. Patients who are sexually active and unwilling to use highly effective contraceptive methods. The following contraceptive methods with a Pearl Index lower than 1% are regarded as highly effective:

    1. Oral hormonal contraception ('pill')
    2. Dermal hormonal contraception
    3. Vaginal hormonal contraception (NuvaRing®)
    4. Contraceptive plaster
    5. Long-acting injectable contraceptives
    6. Implants that release progesterone (Implanon®)
    7. Tubal ligation (female sterilisation)
    8. Intrauterine devices that release hormones (hormone spiral)
    9. Double barrier methods This means that the following are not regarded as safe: condom plus spermicide, simple barrier methods (vaginal pessaries, condom, and female condoms), copper spirals, the rhythm method, basal temperature method, and the withdrawal method (coitus interruptus).

    Except: Female patients who are surgically sterilised by hysterectomy or who are expected to be postmenopausal are eligible for this trial. A lack of menstruation of at least 12 months will be considered as a proof to be postmenopausal.

    Men must agree to use a latex condom during sexual contact with females of childbearing potential while participating in this study even if they have undergone a successful vasectomy.

    Patients must abstain from donating blood, semen, or sperm during participation in the study.
11. Simultaneous participation in any other interventional clinical trial within the last 14 days before the start of this trial; simultaneous participation in registry and diagnostic trials is allowed;
12. Patients without legal German language capacity who are unable to understand the nature, significance and consequences of the trial or any other co-existing medical or psychological condition that will preclude participation in the study;
13. Persons who are in a relationship of dependence/employment with the sponsor or the investigator will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study design | 12 months
  Rates of patient recruitment per month, screening failures, drop-out from the trial.
Number of patients who show no relevant increase of nausea | day 1 to day 6
  Number of patients who show no relevant increase of nausea after starting opioid therapy at any of the following 6 days. Nausea scores are assessed on an increasing 11-point numeric rating scale (NRS) from 0 to 10, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity according to the Edmonton Symptom Assessment Schedule (ESAS). Relevant is an increase on this NRS ≥1, which reflects the minimal clinically important difference (MCID) for nausea

SECONDARY OUTCOMES:
Complete response of OINV | day 1 to day 6
  Complete response defined as no emetic episodes, no nausea, no rescue anti-emetic. Comparing Palonosetron treatment with placebo
Time to OINV | day 1 to day 6
  Time to emetic episodes or nausea or rescue antiemetic after randomisation, comparing Palonosetron treatment with placebo
Nausea | day 1 to day 6
  Occurrence and severity of nausea rated by the participants on a 11-point numeric rating scale (NRS), comparing Palonosetron treatment with placebo. Nausea scores are assessed on an increasing 11-point numerical scale from 0 to 10, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity according to the Edmonton Symptom Assessment Schedule (ESAS).
Vomiting | day 1 to day 6
  Occurrence of vomiting, comparing Palonosetron treatment with placebo
Pain control | day 1 to day 6
  Daily opioid intake and pain score rated by the participants on a 11-point numeric rating scale (NRS). Pain scores are assessed on an increasing 11-point numerical scale from 0 to 10, 0 meaning that the symptom is absent and 10 that it is of the worst possible severity according to the Edmonton Symptom Assessment Schedule (ESAS)
Rescue anti-emetics | day 1 to day 6
  The use of rescue anti-emetics, comparing Palonosetron treatment with placebo
Participant's burden by nausea, pain, constipation and headache | day 1 to day 6
  Assessed by a questionnaire: Patients are asked to assign the burden of their symptoms to one of 4 categories: not at all, a little, strongly, extremely strongly
Severity of constipation | day1 and day 6
  Stool consistency and frequency, bowel function index (BFI)
Symptom preferences | day1 and day 6
  Patients were asked to rank 5 possible symptoms (tumor pain, nausea, vomiting, constipation, headache) from their most undesired to their most acceptable symptom. Rated by the participants at day 6 and compared to baseline.
Percentage of participants reporting any grade 3 adverse event (AE) or any serious adverse event (SAE) from patients from the time of the signed ICF to the end of the study. | day 1 to day 6
  An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
  An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity or is a congenital anomaly/birth defect.
Patient satisfaction with the study drug | day 6
  Patients are asked to rate speed of action of the study drug received, the satisfaction with the overall control of nausea and emesis using 4 categories (very satisfied, satisfied, dissatisfied, very dissatisfied) and the and willingness to use the study drug again (yes, no, unknown). Rated by the participants at day 6.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhild Becker, Prof. Dr. med., Study Chair — Clinic for Palliative Care, Medical Center, University of Freiburg, Germany
Locations (1):
- Clinic for Palliative Care, Medical Center, University of Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No